CLINICAL TRIAL: NCT03085966
Title: Study of Autologous Immune Cell Therapy in Combination With the Luteinizing Hormone Releasing Hormone Agonists (LHRH-a) in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: Autologous Immune Cell Therapy in Combination With LHRH-a in Patients With mCRPC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNWK2016-08-04
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: central memory T cell; metastatic castration-resistant prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous immune cell therapy (Experimental): Luteinizing Hormone Releasing Hormone Agonists (LHRH-a) and Autologous dendritic cells (DC) and central memory T cells (Tcm cells)
  Interventions: Biological: autologous immune cell therapy

INTERVENTIONS:
Biological: autologous immune cell therapy — Luteinizing Hormone Releasing Hormone Agonists (LHRH-a) and Autologous dendritic cells (DC) and central memory T cells (Tcm cells)

SUMMARY:
Study of autologous immune cell therapy in combination with the luteinizing hormone releasing hormone agonists (LHRH-a) in patients with metastatic castration-resistant prostate cancer

DETAILED DESCRIPTION:
Autologous dendritic cells (DC) are known to activate other immune cells, such as central memory T cells (Tcm cells), that are able to mount an attack against cancer cells. The purpose of this study is to evaluate the feasibility, safety and efficacy of patients' own immune cells combined with the luteinizing hormone releasing hormone agonists (LHRH-a) for treatment of metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males age ≥ 18 years；
* Subjects who understand and sign the consent form for this study；
* Metastatic， castrate resistant, histologically confirmed prostate cancer；
* PSA> 5ng / ml；
* Serum testosterone ≤ 17nmol / L (50ng / dl)；
* Expected survival time of at least 24 months；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Subjects did not receive chemotherapy, radiation therapy, surgery and other treatment within 4 weeks；

Exclusion Criteria:

* The subject has an allergic history of medicine or food；
* The patient with more serious heart disease, including but not limited to myocardial infarction, cardiomyopathy, valvular disease, malignant arrhythmia；
* Hb <9.0 g / 100ml, WBC <3 ×10^9/ L, LY <1.0 x10^9/ L, platelet <100,000 / mm3；
* Patients with immune disease or auto-immune disease (such as Multiple sclerosis, systemic lupus erythematosus，rheumatoid arthritis and inflammatory bowel disease, vitiligo )；
* The subject has uncontrolled or hard-to-control diseases of liver, or kidney system；
* Patient with visceral metastases, pathological fractures, spinal cord compression symptoms；
* Severe pain associated with bone metastases (VAS score ≧ 4 points)；
* Patient has received immunotherapy (including but not limited to PD-1 / PDL-1, etc.)；
* patient with irregular hemorrhagic disease；
* Subject is HIV, hepatitis B virus, hepatitis C virus, Treponema pallidum infection；
* Subject has uncontrollable seizures, or because of mental loss of self-knowledge and so on；
* The subject has an history of other malignant tumor；
* The patient had drug abuse, drug abuse, and long history of alcoholism in the 12 years prior to this trial；
* The subject has participated in any other clinical trial in the 3 months prior to this trial；
* The subject has any other unsuitable or adverse condition to be determined by the investigator.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-10-27 (Estimated); Study Completion 2019-12-27 (Estimated)

PRIMARY OUTCOMES:
AE and SAE | 24 months
  Incidences of adverse events or serious adverse events

SECONDARY OUTCOMES:
OS | 24 months
  Overall survival
PFS | 24 months
  Progression-Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai Shi, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided